CLINICAL TRIAL: NCT06184555
Title: Primary Tumor Sidedness Associated With Clinical Characteristic and Postoperative Outcomes in Colon Cancer: a Propensity Score Matching Study
Status: Completed | Type: Observational
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Wan-Hsiang Hu, Attending physician, Chang Gung Memorial Hospital
Other Study IDs: 20231214NSQIP
Record Dates: First submitted 2023-12-14; First posted 2023-12-28 (Actual); Last update posted 2023-12-28 (Actual); Status verified 2013-12

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- colorectal cancer: colectomy

SUMMARY:
Background: Recent investigations have suggested that sidedness is associated with the prognosis of colon cancer patients. The role of sidedness in surgical outcome is unclear. The aim of this study was to investigate the different clinical characteristics and associated postoperative outcomes of sidedness in colon cancer.

Materials and methods: This is a retrospective study using the multi-institutional, nationally validated database of the American College of Surgeons-National Surgical Quality Improvement Program (ACS-NSQIP) from 2009 to 2013. Sidedness groups including right sided and left sided colon cancer were created according to the associated diagnosis and procedure codes. Postoperative mortality, morbidity, overall complication, and length of total hospital stay were analyzed after using a propensity score matching method.

ELIGIBILITY:
Inclusion Criteria:

* colon cancer S/P colectomy

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: colon cancer patients
Sampling Method: Non-Probability Sample
Enrollment: 24436 (Actual)
Dates: Start 2009-01-01 (Actual); Primary Completion 2013-12-31 (Actual); Study Completion 2013-12-31 (Actual)

PRIMARY OUTCOMES:
postoperative complication | one month